CLINICAL TRIAL: NCT01956448
Title: Randomized Clinical Comparison of Biomatrix Flex® and Resolute Integrity® Coronary Stents in Non-selected Patients With Ischemic Heart Disease The SORT OUT VI Study*
Brief Title: SORT-OUT VI - Randomized Clinical Comparison of Biomatrix Flex® and Resolute Integrity®
Acronym: SO VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Biosensors International (Other); Medtronic Cardiovascular (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, DMSc, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110037
Record Dates: First submitted 2012-06-04; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Percutaneous coronary intervention; DES; Angina pectoris; Stent
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug eluting stent (BioMatrix Flex) (Experimental): Device: Percutaneous coronary intervention with implantation of drug eluting stent (BioMatrix Flex)
  Interventions: Device: Drug eluting stent
- Drug eluting stent (Resolute Integrity) (Experimental): Device: Percutaneous intervention with implantation of drug eluting coronary stent (Resolute Integrity)
  Interventions: Device: Drug eluting stent

INTERVENTIONS:
Device: Drug eluting stent — Device: Percutaneous intervention with implantation of drug eluting coronary stent (Resolute Integrity)
  Other Names: BioMatrix Flex - biolimus eluting stent; Resolute - zotarolimus eluting stent

SUMMARY:
To perform a randomized comparison between the BioMatrix Flex™ and the Resolute Integrity® stents in the treatment of unselected patients with ischemic heart disease.

DETAILED DESCRIPTION:
SORT OUT VI is a randomized, multicenter, all-comer, two-arm, non-inferiority trial comparing the Biolimus-eluting Biomatrix Flex and the Zotarolimus-eluting Medtronic Resolute Integrity in treatment of atherosclerotic coronary artery lesions.

Primary Endpoint:

Target lesion failure within 12 months of stent implantation (combination of cardiac death, myocardial infarction (not index procedure related) not related to other than index lesion or target lesion revascularization).

Secondary Endpoints:

Individual components of the primary end point comprised the secondary end points and stent thrombosis rate according to the Academic Research Consortium definition (see protocol for further specification of secondary endpoints).

Clinically driven event detection will be used to avoid study-induced reinterventions. Data on mortality, hospital admission, coronary angiography, repeat percutaneous coronary intervention, and coronary bypass surgery will be obtained for all randomly allocated patients from the following national Danish administrative and healthcare registries: the Civil Registration System; the Western Denmark Heart Registry; the Danish National Registry of Patients, which maintains records on all hospitalizations in Denmark; and the Danish Registry of Causes of Death

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over with chronic stable coronary artery disease or acute coronary syndromes, and at least one coronary artery lesion with more than 50% diameter stenosis, requiring treatment with a drug-eluting stent.

Exclusion Criteria:

* life expectancy of less than one year
* an allergy to aspirin, clopidogrel, ticagrelor, prasugrel, sirolimus, or biolimus
* participation in another randomized trial
* inability to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Device-related combined endpoint | 1,2,3 and 5 years
  Device-related combined endpoint hierarchically:
  cardiac death, non-index procedure related acute myocardial infarction not clearly related to another lesion than the target lesion (new revascularization by PCI or CABG) within 12 months.

SECONDARY OUTCOMES:
Device success rate | 12 months
Procedure success rate | 12 months
Procedure time | 12 months
Fluoroscopy time | 12 months
Amount of contrast | 12 months
Combined endpoint of cardiac death, non-index procedure related acute myocardial infarction, not clearly related to another lesion than target lesion, target lesion revascularisation | 30 days
Target lesion revascularisation | 1,2,3 and 5 years
Death and myocardial infarction | 1 and 12 months
Stent thrombosis | 1,2,3 and 5 years
Device-related combined endpoint hierarchically cardiac death, non-index procedure related AMI, not clearly related to another lesion than target lesion | 2,3 and 5 years
Patient-related combined endpoint hierarchically: all-cause death, non-index procedure related acute myocardial infarction, all new revascularizations | 1,2,3 and 5 years
All-cause death | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ravkilde, MD, Principal Investigator — Aalborg University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Skejby, Aarhus N
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Raungaard B, Christiansen EH, Botker HE, Hansen HS, Ravkilde J, Thuesen L, Aaroe J, Villadsen AB, Terkelsen CJ, Krusell LR, Maeng M, Kristensen SD, Veien KT, Hansen KN, Junker A, Madsen M, Andersen SL, Jensen SE, Jensen LO; SORT OUT VI Investigators. Comparison of Durable-Polymer Zotarolimus-Eluting and Biodegradable-Polymer Biolimus-Eluting Coronary Stents in Patients With Coronary Artery Disease: 3-Year Clinical Outcomes in the Randomized SORT OUT VI Trial. JACC Cardiovasc Interv. 2017 Feb 13;10(3):255-264. doi: 10.1016/j.jcin.2016.11.007. Epub 2017 Jan 18. PMID 28109874
- [Derived] Raungaard B, Jensen LO, Tilsted HH, Christiansen EH, Maeng M, Terkelsen CJ, Krusell LR, Kaltoft A, Kristensen SD, Botker HE, Thuesen L, Aaroe J, Jensen SE, Villadsen AB, Thayssen P, Veien KT, Hansen KN, Junker A, Madsen M, Ravkilde J, Lassen JF; Scandinavian Organization for Randomized Trials with Clinical Outcome (SORT OUT). Zotarolimus-eluting durable-polymer-coated stent versus a biolimus-eluting biodegradable-polymer-coated stent in unselected patients undergoing percutaneous coronary intervention (SORT OUT VI): a randomised non-inferiority trial. Lancet. 2015 Apr 18;385(9977):1527-35. doi: 10.1016/S0140-6736(14)61794-3. Epub 2015 Jan 16. PMID 25601789